CLINICAL TRIAL: NCT00318656
Title: Comparison of the Effects of Rosiglitazone and Glimepiride, Both Given in Combination With Metformin, on 24-Hour Glycemia in Type 2 Diabetes Patients Not Controlled With Metformin Alone. A 3-Month Multicentre, Randomized, Parallel-Group, Open-Label Study.
Brief Title: 24-Hour Glycemia: Rosiglitazone Versus Glimepiride In Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104988; AVAF4003
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Results first posted 2009-03-18 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-04

CONDITIONS: Non-Insulin-Dependent Diabetes Mellitus
Keywords: type 2 diabetes; rosiglitazone; metformin; glimepiride; glycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rosiglitazone-metformin combination; Metformin; glimepiride

INTERVENTIONS:
Drug: rosiglitazone-metformin fixed dose combination
Drug: metformin + glimepiride
  Other Names: rosiglitazone-metformin fixed dose combination

SUMMARY:
A better glycemic control is associated with less complications (cardiac diseases, blindness, etcetera) for type 2 diabetic patients. The objective is to study if rosiglitazone may lead to a more regular glycemic pattern with less hyperglycemia and hypoglycemia episodes than with a sulphonylurea (glimepiride).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 40 to 80 years
* Diagnosis of type 2 diabetes mellitus for at least 6 months
* Body mass index (BMI) ≥25kg/m2
* 7%≥HbA1c ≤ 9% at visit 2
* Treatment with metformin between 1.7g/day and 3g/day for at least 12 weeks prior to visit 1
* Female subjects must be non-pregnant, post-menopausal, surgically sterile or using effective contraceptive measures
* Written informed consent

Exclusion Criteria:

* Use of any oral antidiabetic drug other than metformin within 12 weeks prior to screening
* Significant hypersensitivity to thiazolidinediones and sulfonylureas or compounds with similar chemical structure
* Subjects who have required the use of insulin for glycaemic control at any time in the past or subject with a history of metabolic acidosis including diabetic ketoacidosis
* Subjects with clinically significant ongoing oedema or with a history of oedema in the 12 months prior to visit 1
* Subjects with a history of severe hypoglycaemia
* Anemia defined by haemoglobin concentration <11.0g/dL for males or <10.0g/dL for females
* Renal disease or renal dysfunction, e.g. as suggested by serum creatinine levels ≥135µmol/L in males and ≥110µmol/L in females
* Presence of clinically significant hepatic disease (i.e. ALT, AST, total bilirubin or alkaline phosphatase >2.5 times the upper limit of the normal reference range)
* Congestive heart failure (NYHA class I to IV), unstable or severe angina, recent myocardial infarction
* Subjects with chronic diseases requiring periodic or intermittent treatment with oral or intravenous corticosteroids
* Female who are lactating, pregnant, or planning to become pregnant
* Any clinically significant abnormality identified at screening which in the judgement of the investigator makes the subject unsuitable for inclusion in the study (e.g. physical examination, laboratory test, ECG, ...)
* Use of any investigational agent within 30 days or 5 half-lives (whichever is longer) prior to enrolment in this study
* Active alcohol, drug or medication abuse within the last 6 months or any condition that would indicate the likelihood of poor subject compliance
* Subjects not willing to comply with the procedures described in this protocol.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Monnier L, Colette C, Comenducci A, Vallee D, Dejager S. Add-on therapies to metformin in type 2 diabetes: what modulates the respective decrements in postprandial and basal glucose? Diabetes Technol Ther. 2012 Oct;14(10):943-50. doi: 10.1089/dia.2012.0045. Epub 2012 Jul 9. PMID 22775317

RESULTS

PARTICIPANT FLOW:
Groups:
- Avandamet® (Rosiglitazone/Metformin): Fixed-dose combination will be started at a dose of 4mg/day of Rosiglitazone (RSG) and 2g/day of metformin, i.e. two 1mg/500mg tablets twice daily. After 8 weeks of treatment, the daily dose will be increased to 8mg of RSG and 2g of metformin, i.e. two 2mg/500mg tablets twice daily.
- Glimepiride/Metformin: Metformin will used at a daily dose of 2g, i.e. two 500mg tablet twice daily throughout the study
  Glimepiride will be initiated at a dose of 1mg/day, i.e. half a 2mg tablet od; then, every 2 weeks, the daily dose will be uptitrated up to 4mg/day or until the maximal tolerated dose, using the following pattern:
  * from visit 5 to visit 6: 1mg once a day (half 2mg tablet) before or during breakfast or the first mean meal
  * from visit 6 to visit 7: 2mg once a day (one 2mg tablet) before or during breakfast or the first mean meal
  * from visit 7 to visit 8: 3mg once a day (one and half 2mg tablets) before or during breakfast or the first mean meal
  * from visit 8 onward: 4mg once a day (two 2mg tablet) before or during breakfast or the first mean meal.
Period: Overall Study
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Started | 12 | 11
Completed | 12 | 9 (1 patient received by error avandamet treatment and 1 patient did not receive any treatment.)
Not Completed | 0 | 2
Not completed — Took Avandamet instead of Glim/Met | 0 | 1
Not completed — Did not receive any treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Avandamet® (Rosiglitazone/Metformin): Fixed-dose combination will be started at a dose of 4mg/day of RSG and 2g/day of metformin, i.e. two 1mg/500mg tablets twice daily. After 8 weeks of treatment, the daily dose will be increased to 8mg of RSG and 2g of metformin, i.e. two 2mg/500mg tablets twice daily.
- Total: Total of all reporting groups
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin | Total
Number analyzed (Participants) | 11 | 10 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (10.3) | 62.2 (6.6) | 60.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 8 | 14
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — BMI: A key index for relating a person's body weight to their height. The body mass index (BMI) is a person's weight in kilograms (kg) divided by their height in meters (m) squared.
  kg/m² | 32.2 (6.6) | 30.1 (4.8) | 31.2 (5.8)
HbA1c [Mean (Standard Deviation); unit: percentage] — HbA1c reflects the mean level of glycaemia over time.
  percentage | 7.8 (0.51) | 7.8 (0.52) | 7.8 (0.50)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Hyperglycaemia (>126 mg/dL) in Hours at Baseline Compared to After 12 Weeks on Treatment
Description: Continuous Glycemic Monitoring System, Medtronic (CGMS®) System Gold downloads data to a computer for evaluation of glucose variations.
Time Frame: Baseline and 12 weeks
Population: ITT (randomized): This Intent-to-treat (ITT) population included all subjects who had been randomised, who had received at least one dose of study medication, and for whom at least one efficacy criteria on treatment period was available. The ITT population was the primary population for the efficacy analysis.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Hours
  Baseline | 17.31 (6.25) | 17.53 (6.84)
  12 weeks | 15.30 (6.10) | 10.83 (6.06)
Statistical Analysis 1: Comparison: Avandamet® (Rosiglitazone/Metformin) vs Glimepiride/Metformin; Statistical analysis was based off of week 12 results; Test type: Superiority or Other; p = 0.064, ANCOVA; Analysis of covariance (ANCOVA); Mean Difference (Net) = 5.02, 95% CI [-0.32 to 10.36], Standard Error of Mean 2.49 — Mean Difference =(Rosiglitazone + Met) - (Glimepiride+Met)

2. Primary Outcome: Episodes of Hyperglycaemia (>126 mg/dL) at Baseline Compared to After 12 Weeks on Treatment
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Episodes
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Episodes
  Baseline | 3.91 (2.03) | 4.05 (2.51)
  12 weeks | 5.36 (2.67) | 5.90 (3.01)
Statistical Analysis 1: Comparison: Avandamet® (Rosiglitazone/Metformin) vs Glimepiride/Metformin; Statistical analysis was based off of week 12 results; Test type: Superiority or Other; p = 0.923, ANCOVA — P value von elteren (adjusted on sex); Mean Difference (Net) = -0.26, 95% CI [-3.37 to 2.85], Standard Error of Mean 1.45 — Mean Difference =(Rosiglitazone + Met) - (Glimepiride+Met)

3. Secondary Outcome: Duration of Severe Hyperglycaemia (>150 mg/dL) in Hours at Baseline Compared to After 12 Weeks on Treatment
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Hours
  Baseline | 11.28 (8.67) | 12.35 (7.13)
  12 weeks | 6.39 (5.30) | 4.23 (5.32)

4. Secondary Outcome: Episodes of Severe Hyperglycaemia (>150 mg/dL) at Baseline Compared to After 12 Weeks on Treatment
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Episodes
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Episodes
  Baseline | 4.00 (1.95) | 3.55 (1.34)
  12 weeks | 5.00 (2.98) | 2.95 (2.83)

5. Secondary Outcome: Duration of Hypoglycaemia (<80 mg/dL) in Hours at Baseline Compared to After 12 Weeks on Treatment
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Hours
  Baseline | 0.85 (1.54) | 0.24 (0.45)
  12 weeks | 0.64 (1.97) | 0.41 (0.80)

6. Secondary Outcome: Episodes of Hypoglycaemia (<80 mg/dL) at Baseline Compared to After 12 Weeks on Treatment
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Episodes
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Episodes
  Baseline | 0.64 (0.87) | 0.30 (0.63)
  12 weeks | 0.50 (1.36) | 0.80 (1.60)

7. Secondary Outcome: Duration of Hypoglycaemia (<60 mg/dL) in Hours at Baseline Compared to After 12 Weeks on Treatment
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Hours
  Baseline | 0.51 (1.06) | 0 (0)
  12 weeks | 0.14 (0.47) | 0.08 (0.26)

8. Secondary Outcome: Episodes of Hypoglycaemia (<60 mg/dL) at Baseline Compared to After 12 Weeks on Treatment
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Episodes
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Episodes
  Baseline | 0.50 (1.02) | 0 (0)
  12 weeks | 0.14 (0.45) | 0.1 (0.32)

9. Secondary Outcome: HbA1c (Glycosylated Hemoglobin)
Description: Uncontrolled HbA1c>8.5%. HbA1c and fasting blood glucose taken at hospital
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
Percentage
  Baseline | 7.8 (0.65) | 7.7 (0.50)
  12 weeks | 7.4 (0.62) | 7.1 (0.79)

10. Secondary Outcome: 8-Iso Prostaglandin F2α (8-iso PGF2α) Excretion Rate
Description: 8-Iso Prostaglandin F2α (8-iso PGF2α) excretion rate measured during the 24 hours preceding the CGM system removal. The nocturnal glycemia measured by CGM system will be defined as the average of glycemic values collected between midnight and breakfast time.
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
pg/mL
  Baseline | 361.9 (207.53) | 325.1 (148.2)
  12 weeks | 373.5 (180.15) | 320.4 (84.74)

11. Secondary Outcome: Glycaemia According to CGMS (Nocturnal), mg/dL
Description: Continuous Glycemic Monitoring System, Medtronic (CGMS®) System Gold downloads data to a computer for evaluation of glucose variations.The nocturnal glycemia measured by CGM system will be defined as the average of glycemic values collected between midnight and breakfast time.
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
mg/dL
  Baseline | 148.4 (42.94) | 140.4 (30.18)
  12 weeks | 130.2 (21.97) | 126.3 (21.76)

12. Secondary Outcome: Glycaemia According to CGMS (Diurnal), mg/dL
Description: Continuous Glycemic Monitoring System, Medtronic (CGMS®) System Gold downloads data to a computer for evaluation of glucose variations.The diurnal glycemia measured by CGM system will be the average of glycemic values recorded between breakfast time and midnight.
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
mg/dL
  Baseline | 162.1 (43.1) | 158.7 (27.40)
  12 weeks | 139.1 (15.23) | 130.13 (21.17)

13. Secondary Outcome: Glycaemia According to CGMS (Dawn), mg/dL
Description: Continuous Glycemic Monitoring System, Medtronic (CGMS®) System Gold downloads data to a computer for evaluation of glucose variations.The glycemia "at dawn" measured by CGM system will be defined as the average of glycemic values recorded between 4 AM and breakfast time.
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
mg/dL
  Baseline | 145.0 (37.23) | 138.6 (23.44)
  12 weeks | 130.6 (21.31) | 124.7 (20.26)

14. Secondary Outcome: Glycaemia According to CGMS (Total Area Under the Curve (AUC) for Values Above 1 mg/dL), mg/dL
Description: Continuous Glycemic Monitoring System, Medtronic (CGMS®) System Gold downloads data to a computer for evaluation of glucose variations. The concentrations of glucose will be assessed from the AUC calculations on glycaemic values measured by CGM system.
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
mg/dL
  Baseline | 1428.2 (971.3) | 1293.1 (636.3)
  12 weeks | 891.4 (342.4) | 717.7 (460.6)

15. Secondary Outcome: Glycaemia According to CGMS (Postprandial Incremental AUC or Values Above 1 mg/dL), mg/dL
Description: as for outcome 14
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
mg/dL
  Baseline | 522.8 (271.6) | 443.0 (157.9)
  12 weeks | 356.9 (138.4) | 362.7 (177.3)

16. Secondary Outcome: Glycaemia According to CGMS (Basal Incremental AUC or Values Above 1 mg/dL), mg/dL
Description: as for outcome 14
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
mg/dL
  Baseline | 905.6 (728.2) | 850.1 (601.2)
  12 weeks | 534.5 (307.5) | 355.0 (338.2)

17. Secondary Outcome: Glycaemia According to CGMS (MAGE), mg/dL
Description: Calculation of the Mean amplitude of glycemic excursion (MAGE) was obtained by measuring the arithmetic mean of the major glucose concentration increases or decreases on days 2 and 3 of glycaemic profile and then averaging results on the two days.
Time Frame: Baseline and 12 weeks
Population: ITT (randomized)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Avandamet® (Rosiglitazone/Metformin) | Glimepiride/Metformin
Number analyzed (Participants) | 11 | 10
mg/dL
  Baseline | 75.1 (22.5) | 61.6 (13.7)
  12 weeks | 44.2 (18.3) | 50.8 (16.4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.